CLINICAL TRIAL: NCT05235906
Title: An Open-label, Single Center, Phase II Study of Surufatinib Combined With Sintilimab in Patients With Advanced Adenocarcinoma of the Gastric or Gastrooesophageal Junction Adneocarcinoma Cancer
Brief Title: A Phase II Clinical Study of Surufatinib Combined With Sintilimab in the Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-G104
Record Dates: First submitted 2022-02-09; First posted 2022-02-11 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib + Sintilimab (Experimental)
  Interventions: Drug: Surufatinib+Sintilimab

INTERVENTIONS:
Drug: Surufatinib+Sintilimab — Surufatinib at a dose of 250mg Qd, with humanized anti-PD-1 monoclonal antibody Sintilimab injected intravenously 200mg per 3 weeks until disease progresses or unacceptable tolerability occurs.

SUMMARY:
The efficacy and safety of the use of Surufatinib in combination with Sintilimab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and voluntarily sign informed consent;
2. Age: 18-75 years old;
3. Patients have histologically or cytologically confirmed advanced or recurrent gastric or gastroesophageal junction adenocarcinoma;
4. NO previous therapy for advanced/metastatic disease of GC/GEJ and CPS≥1;
5. Patients have measurable disease as defined by RECIST 1.1 as determined by investigator;
6. Eastern Cooperative Group (ECOG) performance status of 0 to 2;
7. Has adequate organ function;
8. Expected survival period ≥ 3 months;
9. Patients who not received a blood transfusion within 7 days of registration;
10. Patients have recovered adverse events associated with chemotherapy, radiation and surgical operation as pretreatment to Grade 1 or lower with CTCAE v5.0 excluding stable symptoms (eg alopecia, peripheral sensory neuropathy, skin hyperpigmentation, dysgeusia etc.).
11. Patients capable of taking oral medication;
12. Female of childbearing potential who are negative in a pregnancy test within 7 days before enrollment. Both male and female patients should agree to use an adequate method of contraception (total abstinence, an intrauterine device or hormone releasing system, an contraceptive implant and an oral contraceptive) starting with the first dose of study therapy through 6 months after the last dose of study therapy. Duration will be determined when the subject is assigned to treatment.

Exclusion Criteria:

1. Patients who received prior anticancer treatment within 14 days (or 5 times the half-life time, whichever is shorter) or any investigational agent within 28 days prior to the first dose of study drugs.
2. Patients who have undergone surgical treatment and radiotherapy with in 2 weeks before enrollment.
3. Patients with a history of prior treatment with Lenvatinib or any anti-programmed death 1 (anti-PD-1), anti-programmed ligand death 1 (anti-PD-L1), or anti-programmed ligand death 2 (anti-PD-L2 agent).
4. Patients with symptomatic brain metastasis.
5. Patients with hypertension that is difficult to control (systolic blood pressure ≥150 mmHg and diastolic blood pressure ≥100 mmHg) despite treatment with several hypotensive agents.
6. Those who have received live vaccination within 4 weeks before the start of treatment.
7. Patients with active hepatitis.
8. Patients with a history of human immunodeficiency virus (HIV).
9. Patients were judged unsuitable as subject of this trial by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 12 months
Progression-free survival (PFS) | up to 12 months
Overall survival (OS) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer center of SunYat-sen University, Guangzhou, Guangdong, China